CLINICAL TRIAL: NCT01949454
Title: Fluorometholone 0.1% as Perioperative Adjunct Therapy for Lid-rotation Surgery in Trachomatous Entropion and Trichiasis, Dose-varying Study
Brief Title: Fluorometholone as Ancillary Therapy for TT Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Lions Club International Foundation (Other); Berhan Public Health and Eye Care Consultancy PLC (Other); Grarbet Tehadiso Mahber (Other)
Responsible Party: Principal Investigator, John Kempen, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF1707/UND
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Trichiasis; Trachoma; Bilamellar Tarsal Rotation
Keywords: trachoma; trichiasis; trachomatous trichiasis; bilamellar tarsal rotation; fluorometholone; placebo controlled
MeSH Terms: conditions — Trichiasis; Trachoma | interventions — Fluorometholone; Ophthalmic Solutions; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Fluorometholone 0.1% 1 gtt bid x4weeks (Experimental): Fluorometholone 0.1% 1 drop two times daily for four weeks
  Interventions: Drug: Fluorometholone 0.1% ophthalmic solution
- Artificial Tears 1 gtt bid x4 weeks (Placebo Comparator)
  Interventions: Other: Artificial tears (Placebo)
- Fluorometholone 0.1% 1 gtt qid x 4 weeks (Experimental): Fluorometholone 0.1% 1 drop four times daily for four weeks
  Interventions: Drug: Fluorometholone 0.1% ophthalmic solution
- Artificial Tears 1 gtt qid x4 weeks (Placebo Comparator)
  Interventions: Other: Artificial tears (Placebo)
- Fluorometholone 0.1% 1 gtt qid x 8 weeks (Experimental): Fluorometholone 0.1% 1 drop four times daily for eight weeks
  Interventions: Drug: Fluorometholone 0.1% ophthalmic solution
- Artificial Tears 1 gtt qid x8 weeks (Placebo Comparator)
  Interventions: Other: Artificial tears (Placebo)

INTERVENTIONS:
Drug: Fluorometholone 0.1% ophthalmic solution
  Arms: Fluorometholone 0.1% 1 gtt bid x4weeks; Fluorometholone 0.1% 1 gtt qid x 4 weeks; Fluorometholone 0.1% 1 gtt qid x 8 weeks
Other: Artificial tears (Placebo) — Artificial tears (Placebo)
  Arms: Artificial Tears 1 gtt bid x4 weeks; Artificial Tears 1 gtt qid x4 weeks; Artificial Tears 1 gtt qid x8 weeks

SUMMARY:
The investigators aim to evaluate a new potentially cost-effective approach to improving trichiasis surgery outcomes, perioperative topical anti-inflammatory therapy. The investigators hypothesize that adjunctive topical fluorometholone therapy following trichiasis surgery will reduce the risk of recurrent trichiasis. The rationale for this hypothesis is that interruption of inflammation postoperatively would reduce postoperative scarring, leading to better outcomes. As an initial step toward evaluating this modality, the investigators believe it to be necessary to evaluate topical corticosteroid therapy in a safety-oriented study, for which the investigators also hypothesize that fluorometholone will have a perioperative safety profile acceptable for large-scale programmatic use. Topical corticosteroid therapy is associated with potential risks of cataract induction and intraocular pressure (IOP) elevation in susceptible individuals. Fluorometholone has lower intraocular penetration than alternative corticosteroids, with correspondingly less IOP-raising effect while still having favorable effects on conjunctival inflammation, and is a low-cost generic drug. Its poor delivery of corticosteroid into the eye itself provides an advantage in this setting, as the major side effects of therapy are the result of intraocular effects, and therapy only is needed to the conjunctiva. However, prior to use in a large-scale trial it is sensible to make sure adverse outcomes are not observed in a substantial number of TT patients in a smaller scale trial. Secondary goals of such a trial are to evaluate alternative topical corticosteroid dosing schedules to identify an optimal dosing schedule and to identify any preliminary signals of potential efficacy.

DETAILED DESCRIPTION:
Protocol Title: Fluorometholone 0.1% as Perioperative Adjunct Therapy for Lid-rotation Surgery in Trachomatous Entropion and Trichiasis, Dose-varying Study

Study Design: Randomized, double-masked, dose-ranging study of three dose levels of fluorometholone 0.1% or placebo in one eye of subjects with trachomatous trichiasis (TT) undergoing lid rotation surgery

Primary Study Objective: Evaluate the safety and tolerability of three (3) doses of fluorometholone 0.1% in subjects with trachomatous trichiasis (TT) undergoing lid rotation surgery (Bilamellar Tarsal Rotation)

Secondary Study Objective: Conduct a preliminary assessment of the efficacy of three (3) doses of fluorometholone 0.1% in subjects with trachomatous trichiasis (TT) undergoing lid rotation surgery (Bilamellar Tarsal Rotation)

Number of Subjects: Up to 156 eyes of up to 156 subjects

Study Population: Subjects with trachomatous trichiasis (TT) undergoing lid rotation surgery (Bilamellar Tarsal Rotation)

Test Articles:

1. Fluorometholone 0.1% one drop twice daily for four weeks
2. Placebo one drop twice daily for four weeks
3. Fluorometholone 0.1% one drop four times daily for four weeks
4. Placebo one drop four times daily for four weeks
5. Fluorometholone 0.1% one drop four times daily for eight weeks
6. Placebo one drop four times daily for eight weeks

Visit Schedule: Following trichiasis surgery on Day 0, subjects will return for study visits approximately on Days 14, 28, 56, 90, and 365

Tolerability Parameters:

* Treatment-emergent ocular symptoms/signs
* Discontinuation of drug / treatment because of side effects

Safety Parameters:

* Intraocular pressure elevation ≥30 mm Hg
* Cataract
* Adverse events
* Treatment emergent abnormal ophthalmic findings
* Treatment emergent external examination findings
* Visual acuity

Efficacy Parameters:

* Trichiasis recurrence
* Entropion recurrence
* Trachoma activity grade (to the extent activity can be graded in eyes with severe trachomatous scarring)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more
2. Diagnosis with trachomatous trichiasis
3. Plan for lid rotation surgery (Bilamellar Tarsal Rotation) on at least one upper eyelid
4. LOCS 3 cataract grading is level 3 or less for the nuclear cataract scale, and level 2 or less for the cortical cataract and posterior subcapsular cataract scales.
5. Intraocular pressure between 8-20 mm Hg in the study eye.

Exclusion Criteria:

1. Contraindications to the use of the test articles
2. Known allergy or sensitivity to any medication used in this study, including the study medication or its components (e.g., fluorometholone)
3. Currently taking more than two ocular anti-hypertensive medications in the study eye (prior IOP-lowering surgery is acceptable; combinations of two agents such as Cosopt and Combigan are considered two medications)
4. Glaucoma sufficiently advanced that an intraocular pressure spike potentially would put the patient at substantial risk of vision loss, per study ophthalmologist's judgment.
5. Non-phakic (i.e., pseudophakic or aphakic) study eye (contralateral non-phakic eye is permitted).
6. Other than trachoma, any active ocular infections (bacterial, viral, or fungal), or any active ocular inflammation (e.g., scleritis, iritis).
7. History or diagnosis of ocular herpes or presence of a corneal lesion of suspected herpetic origin; or a diagnosis or suspected diagnosis of ophthalmic mycobacterial infection in either eye.
8. Corneal or scleral thinning in either eye.
9. A severe / serious ocular pathology or medical condition which may preclude study completion.
10. Any condition for which it is anticipated ocular or systemic corticosteroid therapy would be required.
11. Unwilling to discontinue use of contact lenses for the duration of the study (should the unusual circumstance of a trachomatous trichiasis patient who uses contact lenses be encountered)
12. Any significant illness or condition that could, in the investigator's or sub-investigator's opinion, be expected to interfere with the study parameters or study conduct; or put the subject at significant risk
13. For women of childbearing age, currently pregnant and/or breastfeeding, as obtained by self-report (because of concerns about the (programmatic) use of azithromycin in this setting).
14. Cataract in the study eye, defined as LOCS-3 cataract grading is level 3.1 or more for the nuclear cataract scale, or level 2.1 or more for the cortical cataract or posterior subcapsular cataract scales.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety assessments | Within one year of randomization
  Incident cataract is defined as either: 1) a two-step worsening on the nuclear, cortical, and/or posterior subcapsular LOCS-3 scale; or 2) undergoing cataract surgery prior to that point in follow-up.
  Intraocular pressure elevation
  Other dose-limiting toxicity: 1) SAEs (see below) judged as likely related to the treatment by the investigators; 2) vision-threatening non-trachoma infections, e.g., corneal ulcer; 3) anaphylaxis or other events requiring immediate resuscitation; or 4) when the clinician-investigators determine that other AEs observed in a subject would make future applications of the treatment contraindicated on the basis of side effects.

SECONDARY OUTCOMES:
Recurrence of trichiasis in the study eye | Within one year of randomization
  Lashes touching the globe or cornea

OTHER OUTCOMES:
Treatment-emergent ocular symptoms/signs | Within 4-8 weeks
  Within the period of randomized treatment (either 4 or 8 weeks from randomization)
Discontinuation of drug / treatment because of side effects | Within 4-8 weeks of randomization
  During the period of treatment (either 4 or 8 weeks after randomization)
Other adverse events | Within 1 year
Visual acuity | Within 1 year
  Changes from baseline. Changes could either be favorable or unfavorable.
Entropion recurrence | Within 1 year
  Among cases with entropion at baseline, the incidence of entropion recurrence.
Trachoma activity grade | Within 1 year
  WHO trachoma activity grade (to the extent activity can be graded in eyes with severe trachomatous scarring)

CONTACTS AND LOCATIONS:
Overall Officials: John H Kempen, MD MPH PhD, Principal Investigator — University of Pennsylvania; Wondu Alemayehu, MD, MPH, Principal Investigator — Berhan Public Health & Eye Care Consultancy PLC
Locations (1):
- Grarbet Tehadiso Mahber (Grarbet Hospital), Butajīra, Snnpr, Ethiopia